CLINICAL TRIAL: NCT02572713
Title: Systemic Synuclein Sampling Study (S4)
Acronym: S4
Status: Completed | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: Indiana University (Other); University of Iowa (Other); Banner Health (Other); Paracelsus Elena Klinik (Other)
Responsible Party: Principal Investigator, Lana Chahine, MD, Clinical Co-PI, University of Pennsylvania
Other Study IDs: S4-001
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; alpha-synuclein; biomarker
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — ioflupane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biofluid samplings [blood, saliva, and cerebrospinal fluid (CSF)] Tissue samplings (skin, colon, submandibular gland)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Early PD: 20 early PD not requiring dopamine replacement therapy have been enrolled.
  Interventions: Procedure: Biofluid samplings; Procedure: Tissue samplings; Drug: DaTSCAN™
- Moderate PD: 20 moderate PD on dopamine replacement therapy without motor fluctuations have been enrolled.
  Interventions: Procedure: Biofluid samplings; Procedure: Tissue samplings; Drug: DaTSCAN™
- Advanced PD: 21 advanced PD with motor fluctuations have been enrolled.
  Interventions: Procedure: Biofluid samplings; Procedure: Tissue samplings; Drug: DaTSCAN™
- Healthy Controls: 21 healthy controls have been enrolled.
  Interventions: Procedure: Biofluid samplings; Procedure: Tissue samplings; Drug: DaTSCAN™

INTERVENTIONS:
Procedure: Biofluid samplings — Biofluid samplings (blood, saliva, and cerebrospinal fluid (CSF)
Procedure: Tissue samplings — Tissue samplings (skin, colon, submandibular gland)
Drug: DaTSCAN™
  Other Names: ioflupane-123I

SUMMARY:
The purpose of this study is to measure alpha-synuclein in peripheral body tissues and fluids in Parkinson's disease (PD). This may help in developing better treatments for PD patients in the future.

DETAILED DESCRIPTION:
This is a multi-center, cross-sectional, observational study to evaluate α-syn pathology in multiple tissues and biofluids in individual subjects with PD and HC at a single time point.

ELIGIBILITY:
Inclusion Criteria (PD subjects):

* Male or female age 40 or older at the time of PD diagnosis.
* Clinical diagnosis of PD based on bradykinesia plus one of the following: rest tremor or rigidity.
* DAT deficit at screening based on visual interpretation of DaTSCAN™ imaging.
* PD subjects will need to fall into one of the following stages:

  * Early untreated PD not requiring dopamine replacement medication (anticholinergics, MAO-B inhibitors and amantadine permitted), Hoehn and Yahr 1-2, < 2 years from diagnosis.
  * Moderate PD responsive and currently treated with dopamine replacement therapy without evidence of motor fluctuations or dyskinesias.
  * Advanced PD with motor fluctuations or dyskinesias, > 5 years from diagnosis.
* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* Willing and able to comply with scheduled visits, required study procedures and laboratory tests.

Inclusion Criteria (HC subjects):

* Male or female age 50 or older at the time of the screening visit
* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* Willing and able to comply with scheduled visits, required study procedures and laboratory tests.

Exclusion Criteria (all subjects):

* Has a history of cancer (other than basal and squamous cell skin cancers), autoimmune disorder, liver disease, or other hematological disorder within the past 5 years.
* Current treatment with anticoagulants (e.g., Coumadin, heparin) that would preclude safe completion of the lumbar puncture (LP) and tissue biopsy procedures.
* Current treatment with an antiplatelet agent (Plavix or aspirin >325 mg/day).
* Has a diagnosis of diabetes mellitus requiring either an oral agent or insulin therapy.
* A bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Has received botulinum toxin injections to the submandibular gland within the past year.
* Has a condition that precludes safe performance of routine LP, such as prohibitive lumbar spinal disease.
* Has a condition that precludes the safe performance of the flexible sigmoidoscopy procedure or may interfere with obtaining evaluable colonic tissue biopsies, including a prior colonoscopy with significant findings (e.g. polyp with a positive finding, ulcerative colitis, Crohn's disease, inflammatory disease).
* Has a condition that precludes the safe performance of the submandibular gland procedure or may interfere with obtaining evaluable submandibular tissue biopsies, including any previous or active significant disease affecting the submandibular gland (e.g. inflammatory disease, infection, tumor).
* Has a condition that precludes the safe performance of the skin punch biopsy procedure or may interfere with obtaining evaluable skin tissue biopsies, including any previous or active significant dermatological disease (e.g. previous biopsy with any of the following findings: inflammatory disease, scar tissue, psoriasis, keloid formation, skin cancer).
* Any other medical or psychiatric condition or laboratory abnormality, which in the opinion of the Site Investigator would preclude participation.
* Use of investigational drugs or devices within 30 days prior to the screening visit.

Exclusion criteria (PD subjects):

* Has other significant neurological disorders (clinically significant stroke, brain tumor, hydrocephalus, epilepsy, other neurodegenerative disorders, encephalitis, repeated head trauma, polyneuropathy).
* Has significant autonomic dysfunction (symptomatic orthostasis, hypotension or urinary incontinence) suggestive of an atypical parkinsonism.
* Has atypical features of parkinsonism including but not limited to supranuclear gaze palsy, early recurrent falls, corticospinal track abnormalities, cerebellar abnormalities, significant cognitive dysfunction.

Exclusion criteria (HC subjects):

* Has a family history of PD in any first-degree relative.
* Has a significant neurological disorder (a neurodegenerative condition, clinically significant stroke, brain tumor, hydrocephalus, epilepsy, other neurodegenerative disorders, encephalitis, repeated head trauma, polyneuropathy).
* Has a Montreal Cognitive Assessment (MoCA) score of less than 26.
* Has a diagnosis of REM sleep behavior disorder.
* Has a primary dystonia, restless legs syndrome, essential tremor, or other movement disorder.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited through patient care clinics, physician referrals, and by reaching out to the community (e.g. PD-affiliated groups).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
α-syn levels in blood | 24 months
  Blood will be analyzed using the most optimal, currently available, quantitative assays. The outcome will be expressed as a concentration of α-syn levels.
α-syn levels in saliva | 24 months
  Saliva will be analyzed using the most optimal, currently available, quantitative assays. The outcome will be expressed as a concentration of α-syn levels.
α-syn levels in CSF | 24 months
  CSF will be analyzed using the most optimal, currently available, quantitative assays. The outcome will be expressed as a concentration of α-syn levels.
α-syn deposits in skin | 24 months
  α-syn burden in skin biopsies will be expressed as 1) simply positive or negative, i.e. whether any two slides are positive out of all examined 2) by total percentage of slides examined that are positive 3) by site of highest density of positive α-syn fibers.
α-syn deposits in submandibular gland | 24 months
  α-syn burden in the submandibular tissue will be expressed as 1) simply positive or negative, i.e. whether any two slides are positive out of all examined 2) by total percentage of slides examined that are positive 3) by site of highest density of positive α-syn fibers.
α-syn deposits in colon | 24 months
  α-syn burden in the colon tissue will be expressed as 1) simply positive or negative, i.e. whether any two slides are positive out of all examined 2) by total percentage of slides examined that are positive 3) by site of highest density of positive α-syn fibers.

CONTACTS AND LOCATIONS:
Overall Officials: Lana Chahine, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Toronto Western Hospital Movement Disorders Centre, Toronto, Ontario, Canada